CLINICAL TRIAL: NCT05511545
Title: The Effect of Training Given to Patients Who Underwent Ureteroscopy With Double-J Stent Placement on Anxiety Before and After Surgery and Readiness for Discharge
Brief Title: The Effect of Education Given to Patients on Pre- and Post-operative Anxiety and Preparation for Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muazzez Merve TORAMAN, Research Assistant, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Muazzez
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Kidney Calculi
Keywords: anxiety, double j stent, nurse, education, ureteroscopy
MeSH Terms: conditions — Kidney Calculi; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Education Booklet (Experimental): One day before surgery:
  The patients in the training group were informed about the study one day before the operation and their verbal and written consents were obtained. Afterwards, the Descriptive Information Form, the State-Trait Anxiety Inventory, and the Surgery-Specific Anxiety Inventory were administered. A training booklet was prepared by the researchers in line with the recommendations of the European Association of Urology and the relevant literature. The training took an average of 25-30 minutes. Afterwards, the questions of the patients were answered and the training booklet was given to the patient.The scales were reapplied on the morning of the surgery.
  Before discharge, the State Anxiety Scale and the Readiness to Discharge Scale-Patient Self-Assessment Form were administered. Then, the Adult Patient Discharge Readiness Scale-Nurse Evaluation Short Form was filled by the clinical nurse caring for the patient.
  Interventions: Other: Patient Education Booklet

INTERVENTIONS:
Other: Patient Education Booklet — Excretory system organs, signs and symptoms to be seen in kidney and ureteral stones, treatment methods, ureteroscopy procedure, what to do before and on the morning of surgery, and surgery, using the training booklet prepared by the researchers in line with the recommendations of the European Association of Urology and the relevant literature. An average of 25-30 minutes of training was given in the patient's room in an encouraging language, allowing the patient to ask questions about the situations he would encounter in the clinic after the surgery. She started asking questions she didn't understand. Afterwards, the questions of the patients were answered and the patient was given a training booklet.

SUMMARY:
The data of the randomized controlled experimental research were collected at Atatürk University Health Application and Research Hospital Urology Clinics between November 2021 and May 2022. The study sample consisted of 122 patients (61 in the training group, 61 in the control group) who were selected by the simple random sampling method and met the research inclusion criteria.

DETAILED DESCRIPTION:
Ureteroscopy (URS) is an up-to-date method that is widely used in the diagnosis and treatment of ureteral diseases. Apart from the diagnostic purposes of URS, the most common use is to intervene in ureteral stones. The vast majority of ureteral stones are treated endoscopically. A Double-J (DJ) stent is often placed after ureteroscopy. The purpose of the stent is to prevent obstruction, renal colic, and deterioration of renal function. The fact that the DJ stent will remain in the patient for a certain period of time (approximately 3-4 weeks) causes anxiety in the patient. However, approximately 80% of patients with DJ stent implantation have urinary system symptoms that impair their quality of life. Frequent urination (50-60%), sudden urge to urinate (57-60%), pain on urination (40%), incomplete evacuation (76%), flank pain (19-32%), suprapubic pain (30%) , incontinence and hematuria (25%) are the symptoms seen. Patients with DJ stent implanted after ureteroscopy surgery need more information, support, explanation and help to cope with the effects of these symptoms in the clinic and at home. In this context, it is important to provide an individualized and comprehensive education that includes the home care process before and after the URS. It has been determined in the literature that training before surgery reduces anxiety, pain level, complication and depression rates, and increases patient satisfaction in the postoperative period. No study has been found in the literature examining the effects of education given to patients with URS on their post-operative anxiety and readiness for discharge. In this context, this study will provide evidence-based data to the literature by investigating the effects of training given to patients with URS and DJ stent implantation on pre- and postoperative anxiety and readiness for discharge.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research and volunteering,
* Those between the ages of 18-65,
* Having URS surgery for the first time due to stone and temporary DJ stent placed,
* Patients whose cognitive level scales were suitable for application were included in the study.

Exclusion Criteria:

* Having URS surgery for non-stone causes,
* Permanent stent placed,
* Leaving work voluntarily,
* Patients with major hearing and vision problems were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety İnventory (STAI-I, STAI-II) | up to 24 hours
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Owner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
Surgery Specific Anxiety Scale | up to 24 hours
  This scale was developed in Turkish by Karancı and Dirik in 2003 to measure the pre- and postoperative anxiety of surgical patients. It consists of 10 items in total. Each item is rated on a 5-point Likert-type scale. The surgery-specific anxiety score is obtained by summing the responses to all items. The minimum score that can be obtained from the scale is 10, and the maximum score is 50.
Readiness for Hospital Discharge Scale for Adult Patients-Short Form and Readiness for Hospital Discharge Scale- Adult-Nurse Assesment Short Form | up to 24 hours
  The scale developed by Weiss et al. in 2006 was used by Kaya et al. It was adapted to Turkish in 2018 and has parallel questions with the nurse version, and has a 10-point Likert-type evaluation. The scale, in which the patients' readiness for discharge is evaluated by themselves, consists of eight items and four sub-dimensions. Eight questions in the scale are evaluated with scores between 0-10, from the lowest to the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Muazzez Merve TORAMAN, Principal Investigator — Ataturk University
Locations (2):
- Turkey (Türkiye) (2):
  - Muazzez Merve TORAMAN, Erzurum, Palandöken
  - Muazzez Merve TORAMAN, Erzurum